CLINICAL TRIAL: NCT01584778
Title: The Serum Eosinophil Cationic Protein Levels in Behçet's Disease and Its Relation to the Clinical Activity
Brief Title: Behçet's Disease and Eosinophil Cationic Protein
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Didem Arslan Tas, Dr. Didem Arslan Tas, Cukurova University
Other Study IDs: TF.00.U.32.
Record Dates: First submitted 2012-04-24; First posted 2012-04-25 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Behçet's Disease
Keywords: Behçet's disease; Eosinophil cationic protein; Eosinophils
MeSH Terms: conditions — Behcet Syndrome | interventions — Eosinophil Cationic Protein

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Behçet patients
  Interventions: Other: eosinophil cationic protein
- Healthy controls
  Interventions: Other: eosinophil cationic protein
- Allergic rhinitis (diseased) controls
  Interventions: Other: eosinophil cationic protein

INTERVENTIONS:
Other: eosinophil cationic protein — Serum eosinophil cationic protein levels
  Other Names: ECP

SUMMARY:
Eosinophil cationic protein (ECP) is a matrix protein of eosinophils and has been reported to reflect eosinophil activity. Few studies have examined the role of eosinophils in the pathogenesis of Behçet's disease. The purpose of the present study is to investigate the serum ECP levels in BD and its relation to clinical activity.

DETAILED DESCRIPTION:
Behçet's disease (BD) is a systemic vasculitis, characterized by recurrent oral aphthae, genital ulcers, uveitis, skin lesions, arthritis, gastrointestinal and neurologic manifestations. There has been a growing interest in research on the pathogenesis of the disease. Eosinophils has been implicated in the vascular injury associated with several vasculitis syndromes like Churg Strauss syndrome, temporal arteritis and Henoch-Schonlein purpura. In Behçet patients, serum IgE and eosinophils have been reported to be comparable with the controls but eosinophil activity has not been studied extensively. Eosinophil cationic protein (ECP) is a matrix protein of specific granules of eosinophils with considerable capacity to damage tissue and cells and has been reported to reflect eosinophil activity. Increased serum levels of ECP has been reported in patients with seasonal allergic rhinitis. Several immunomodulatory features of ECP has been reported, such as inhibition of the proliferative T-lymphocyte response to antigen, immunoglobulin production, proliferation of plasma cell lines and upregulation of ICAM-1. Procoagulant effects of ECP has also been reported. The present study was conducted in patients without usage of any confounding drugs that can effect serum ECP levels. The purpose of this study was to investigate the serum ECP levels in BD and its relation to the clinical activity.

Forty-seven consecutive patients with BD (22 active, 25 inactive) meeting International Study Group Criteria , 21 age and sex matched patients with allergic rhinitis and 21 apparently healthy controls were evaluated prospectively in Rheumatology-Immunology Outpatient Clinic. Clinical activity was defined according to the criteria proposed by "Behcet's Disease Research Committee of Japan" . Activity scoring was made according to the "Behçet's Disease Research Committee of Japan" which was proposed in 1994. Organ involvements of the patients were summarized.

Patients on corticosteroids or immunosuppressives were excluded. Colchicine was stopped 10 days prior to the blood collection in inactive patients. Blood was drawn from the active patients before starting treatment. Cases with any allergy history or parasitosis were excluded.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive Behçet patients who gave the written informed consent were included.

Exclusion Criteria:

* Patients on corticosteroids or immunosuppressives were excluded.Cases with any allergy history or parasitosis were excluded.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive Behçet patients of the outpatient clinic of the Rheumatology-Immunology Department of University Hospital
Sampling Method: Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2002-01; Primary Completion 2002-12 (Actual); Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hüseyin TE Ozer, Assoc. Prof., Study Chair — Cukurova University, Faculty of Medicine, Rheumatology-Immunology Department; Eren Erken, Prof. Dr., Study Director — Cukurova University, Faculty of Medicine, Rheumatology-Immunology Department
Locations (1):
- Cukurova University, Faculty of Medicine, Rheumatology-Immunology Department, Adana, Turkey (Türkiye)